CLINICAL TRIAL: NCT07261852
Title: Effects of Muscle Strength Training in Lower Limb Amputee Patients
Brief Title: Muscle Strength Training in Lower Limb Amputee Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Gabriela Dell Elce, principal investigator, University of Gran Rosario
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 619/2024
Record Dates: First submitted 2025-09-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Lower Limb Amputation
Keywords: amputees; quality of life; funcionality; muscle strength; movility; endurance training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle strength training (Experimental): Strength training lasts six weeks, during which submaximal strength percentages ranging from 75% to 90% are worked on.
  It is performed three times a week and follows a protocol consisting of progressive exercises for the large functional muscle groups relevant to the population being trained.
  Interventions: Other: Muscle strengh training
- Endurance training (Active Comparator): Resistance training will be carried out for 6 weeks, 3 times a week, with exercises prescribed by a protocol with training characteristics defined by bibliography found in the ACSM.
  Interventions: Other: Resistence training

INTERVENTIONS:
Other: Muscle strengh training — Strength training lasts six weeks, during which submaximal strength percentages ranging from 75% to 90% are worked on.
  It is performed three times a week and follows a protocol consisting of progressive exercises for the large functional muscle groups relevant to the population being trained.
  Arms: Muscle strength training
Other: Resistence training — Resistance training will be carried out for 6 weeks, 3 times a week, with exercises prescribed by a protocol with training characteristics defined by bibliography found in the ACSM.
  Arms: Endurance training

SUMMARY:
This study is a clinical trial that evaluates the best treatment option using a strength training protocol and an endurance training protocol in patients with lower limb amputations who use prostheses. The protocol consists of 6 weeks of strength training and 6 weeks of endurance training, with a 1-month washout period between the two.

DETAILED DESCRIPTION:
The assessments in this study focus primarily on strength, using a dynamometer and the 5 RM, functionality, using the AMP scale, mobility, using the TugTest, quality of life, using the WHOQOL-BREF, and perception of change, using the GROC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral lower limb amputation
* Transtibial and/or transfemoral amputation
* Prosthetized
* Aged 18 to 75 years
* Who sign the informed consent form

Exclusion Criteria:

* That they are unable to complete the initial assessment
* That they undergo further secondary training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Funcionality | day 1, day 18 (last day of week 6), day 1 (after the wash out) and day 24.
  It is assessed using the TUG test, which requires patients to get up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down again. Patients will receive the following instructions: "Get up on the word 'go,' walk to the tape, turn around, walk back to the chair, and sit down."
Changes in quality of life | day 1, day 18 (last day of week 6), day 1 (after the wash out) and day 24.
  It is assessed using a self-administered questionnaire called WHOQOL-BREF, which provides a profile of the person's perceived quality of life.

SECONDARY OUTCOMES:
Changes in Maximum isometric muscle strength | day 1, day 18 (last day of week 6), day 1 (after the wash out) and day 24.
  It is evaluated using a dynamometer, in which three measurements are taken for each designated movement and the average of the maximum force and peak force is calculated.
Changes on Movility | day 1, day 18 (last day of week 6), day 1 (after the wash out) and day 24.
  It is assessed using the AMP functional rating scale (amputee mobility predictor).
Change in Global percepcion of change | assessments were performed at the end each protocol. day 18 and day 24
  It is an assessment carried out using the Groc scale, which evaluates changes in perception.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro S Barone, Study Director — Ugr

IPD SHARING:
Plan to Share IPD: Yes
If necessary or required, informed consent and data analysis will be shared.
Supporting Information: SAP, ICF